CLINICAL TRIAL: NCT05984576
Title: Radiotherapy & Total Neoadjuvant Therapy for Recurrent Rectal Cancer in Previously Irradiated Patients, an Italian Association for Radiotherapy and Clinical Oncology (AIRO)-GI Platform: a Multi-centre Prospective Observational Study
Acronym: RETRY
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, GAMBACORTA MARIA ANTONIETTA, Professor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 5579
Record Dates: First submitted 2023-05-26; First posted 2023-08-09 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Rectal Neoplasm
Keywords: Radiotherapy; Reirradiation; Recurrent Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms | interventions — Re-Irradiation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: Reirradiation — Reirradiation recurrent rectal cancer

SUMMARY:
The introduction of neoadjuvant chemoradiation therapy (CRT) and the use of advanced surgical techniques have led to a reduction in mortality and recurrence rates for rectal cancer, the rate of which currently stands at 4-8%. Complete cytoreduction (achieving R0) of local recurrence is the main factor correlating with survival, but surgery can often be very complex because of the change in anatomical planes caused by previous surgery. Reirradiation of the recurrence may increase the rate of optimal resection (R0) and may palliate symptoms in unresectable disease. It is a very complex procedure, because one has to take into account the dose previously received by the organs at risk (OARs) and at the same time be able to deliver an effective dose to the recurrence. However with modern irradiation techniques (VMAT) it is possible to increasingly spare the OARs and deliver adequate doses in this setting as well.

Besides radiotherapy with conventional fractionation, other promising options are stereotactic body radiotherapy (SBRT) with and proton (PT) and carbon ion RT (CIRT). Another topic of interest is chemotherapy intensification (CHT): recent studies of concomitant and neoadjuvant chemotherapy (Total Neoadjuvant Therapy) have shown high rates of antitumour response, however even this option should be evaluated with caution, because it must take into account previous cancer treatments received by the patient.

Based on the evidence reported in the literature, it is reasonable to assume that treatment of local recurrence of rectal cancer should be multimodal, integrating surgical treatment with CHT and RT, using the different technologies available. To this end, proper stratification of patients is necessary in order to target the appropriate therapy according to the type of recurrence and their clinical condition.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old;
* Eastern Cooperative Oncology Group (ECOG) 0-1;
* Adequate hematological function, i.e.:
* Granulocyte count > 1500/µL;
* Hemoglobin level >10 g/dL;
* Platelet count > 100000/µL;
* Alanine aminotransferase (ALT)/aspartate aminotransferase (AST): 7-45 international units (UI)/L.
* Potentially curable Oligo-metastatic disease;
* Life expectancy of more than 24 months;
* Histologically (if feasible) or radiologically MRI (magnetic resonance imaging), if no contraindications, and CT (computed tomography) and/or Positron Emission Tomography scan (PET) proven pelvic local recurrent rectal cancer (LRRC);
* Previous pelvic irradiation > 6 months;
* Availability of the previous treatment plan in DICOM format only (Digital Imaging and COmmunications in Medicine).

Exclusion Criteria:

* Age <18 y.o.;
* Pregnancy or lactating female patients;
* Psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule (those conditions should be discussed with the patient before registration in the trial);
* Important comorbidities (such as: severe cardiac or coagulative disease, moderate or severe restrictive/obstructive lung deficit, severe cognitive impairment, moderate and severe renal and hepatic impairment.
* Refusal to sign written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Recurrent rectal cancer previously irradiated
Sampling Method: Non-Probability Sample
Enrollment: 88 (Estimated)
Dates: Start 2023-06-21 (Actual); Primary Completion 2026-06-05 (Estimated); Study Completion 2031-06-05 (Estimated)

PRIMARY OUTCOMES:
Local control | 8 years
  The primary aim of this study is to investigate whether the combination of total neoadjuvant therapy (TNT) with re-RT could lead to a better Local Control rate in Local recurrent rectal cancer patients previously irradiated.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Gemelli, Rome, Italy

REFERENCES:
- [Derived] Gambacorta MA, Romano A, Caravatta L, Macchia G, Chiloiro G, Galofaro E, Valvo F, Vitolo V, Alterio D, Mantello G. Radiotherapy & total neoadjuvant therapy for recurrent rectal cancer in previously irradiated patients, (RETRY): a multicenter prospective observational study. Radiat Oncol. 2024 Dec 18;19(1):174. doi: 10.1186/s13014-024-02555-x. PMID 39695675